CLINICAL TRIAL: NCT04201041
Title: Trans-gluteal Versus Trans-vaginal Pudendal Nerve Fluoroscopic Guided Pulsed Radiofrequency for Treatment of Superficial Dyspareunia: a Prospective Cohort Study
Brief Title: Pudendal Nerve Fluoroscopic Guided Pulsed Radiofrequency for Treatment of Superficial Dyspareunia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: South Egypt Cancer Institute (Other)
Responsible Party: Principal Investigator, Alaa Ali M. Elzohry, Clinical Professor, South Egypt Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PNB
Record Dates: First submitted 2019-12-11; First posted 2019-12-16 (Actual); Last update posted 2020-04-09 (Actual); Status verified 2020-04

CONDITIONS: Superficial Dyspareunia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- trans-gluteal approach (Active Comparator): received pudendal nerve pulsed radiofrequency through trans-gluteal approach
  Interventions: Procedure: pudendal nerve pulsed radiofrequency
- trans-vaginal approach (Active Comparator): received pudendal nerve pulsed radiofrequency through trans-vaginal approach
  Interventions: Procedure: pudendal nerve pulsed radiofrequency

INTERVENTIONS:
Procedure: pudendal nerve pulsed radiofrequency — received pudendal nerve pulsed radiofrequency through trans-vaginal approach or trans-gluteal approach

SUMMARY:
Superficial dyspareunia represents a major health problem especially for the newly wed couples. Pulsed radiofrequency for pudendal nerve is a non-neurolytic neuromodulatory method that is effective in relief of this type of pain. Objectives: to evaluate the efficacy of bilateral pudendal nerve fluoroscopic guided pulsed radiofrequency in treatment of intractable non-organic dyspareunia, and compare between trans-gluteal and transvaginal approaches regarding patient comfort and satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* women aged between 16 and 46 years and from a near vicinity to our facility to make her available for follow-up

Exclusion Criteria:

* We had excluded women with any abnormality in the transvaginal US guided imagining, or those with any evidence of local gynecological abnormalities on examination. Meanwhile, we had excluded those women with infection at site of injection, coagulopathy or other bleeding diathesis, pre-existing neurologic deficit in the targeted region, those with history of chronic opioid use and women who refused to participate in the study

Ages: 16 Years to 46 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2020-03-20 (Actual); Study Completion 2020-03-25 (Actual)

PRIMARY OUTCOMES:
change in Numerical rating scale | baseline reading -1 day reading-3 days postoperative reading
  0 no pain and 10 maximum pain

CONTACTS AND LOCATIONS:
Overall Officials: Alaa Elzohry, MD, Principal Investigator — South Egypt Cancer Institute
Locations (1):
- South Egypt Cancer Institute, Assiut University, Arab Republic of Egypt, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No